CLINICAL TRIAL: NCT02994511
Title: Cambridge Liquid Biopsy and Tumour Profiling Study for Patients on Experimental Therapeutics Trials
Acronym: CALIBRATE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CCTU- Cancer Theme (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, CCTU- Cancer Theme, Dr Richard Baird, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Other Study IDs: CALIBRATE
Record Dates: First submitted 2016-03-17; First posted 2016-12-16 (Estimated); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Cancer
Keywords: Circulating tumour DNA; ctDNA
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumour samples Blood Samples ctDNA isolated from bloods samples
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will explore the potential of the circulating tumour DNA (ctDNA) as predictive factor of response/resistance to anticancer treatment. The project will involve the collection and study of the archived tumour tissue where available (mandatory), serial blood samples (mandatory) and fresh tumour biopsies (optional) from patients taking part in an early phase clinical trial.

DETAILED DESCRIPTION:
Some patients respond to anti-cancer drugs whilst others do not, despite having tumours with, apparently, similar characteristics such as site of origin. This variability in response can in some cases be explained by the genetic profile of the tumour. Therefore, studying the relationship between the molecular profiles of individual cancers and the response to therapy over time is of crucial importance in drug development. However, this endeavour is hampered by the difficulty in accessing suitable tumour material for analysis. Many patients' tumours are at anatomical sites which make biopsy difficult / hazardous which is in addition to the discomfort of a biopsy procedure. Therefore, this study will explore the potential of the circulating tumour DNA as a predictive factor of response/resistance to anticancer treatment.

For patients recruited to early phase clinical trials of experimental therapies, archival tumour tissue (mandatory), serial blood samples (mandatory) and fresh tumour biopsies (optional) will be collected according to the individual schedule of each clinical trial.

Blood plasma samples will be tested for cell-free and ctDNA levels and genomic profiles, which may include analyses of mutational profiles, copy number variations, translocations, chromosomal rearrangements and/or epigenetic profiles.

Molecular profiling of archival and fresh tumour biopsies will also be carried out to study the correlation with cell-free and ctDNA samples and investigate the potential predictor response/resistance to treatment.

ELIGIBILITY:
Inclusion criteria:

* Histological or cytological confirmation of cancer
* Patient being considered for participation in an experimental therapeutic trials
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow up schedule (such conditions should be discussed with the patient before registration in the study)

Exclusion criteria:

* Age below 18 years old
* Patient not physically and mentally able to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients potentially eligible for early phase experimental therapeutic trials will be invited to take part in this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-12-08 (Actual); Primary Completion 2020-03-30 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of the change in circulating tumor DNA [ctDNA] levels of patients on experimental therapeutic trials. | From baseline to the end of study, defined as 'disease progression or evidence of unacceptable toxicity', whichever comes first, measured at the start of each cycle (cycle = approximately 3 weeks) and CT scan (every 2 cycles), for up to 100 months.
  ctDNA levels will be compared to clinical, pathological and radiological data to assess relationship to response and progression of cancer.

SECONDARY OUTCOMES:
Acceptability of research sampling | Optional fresh tissue biopsies are planned to be taken at baseline, at the CT scan day for evaluation of response (every 2 cycles (cycle = approximately 3 weeks)) and after disease progression is confirmed, for up to 100 months.
  Acceptability of research tumour biopsies will be assessed by providing a patient with an 'Acceptability Questionnaire' pre and post biopsy.
Safety of tumour biopsies for patients with cancer on experimental therapeutic trials | Assessed at baseline, at the CT scan day for evaluation of response (every 2 cycles (cycle = approximately 3 weeks)) and after disease progression is confirmed, for up to 100 months.
  Serious Adverse events at least possibly related to the research biopsy procedure will be collected prospectively. In addition, information related to the medical history and biopsy procedure will be recorded at the different time points.
Gene Mutation profiles in ctDNA and tumour biopsies (where available) over time for patients with cancer on experimental therapeutic trials | From baseline, at the time points specified in Outcomes 1 and 2, until the end of study, defined as 'disease progression or evidence of unacceptable toxicity', for up to 100 months.
  Gene mutation profiles will be compared to clinical, pathological and radiological data to assess relationship to response and progression of cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Baird, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom